CLINICAL TRIAL: NCT06822179
Title: Effectiveness of a Personalized In-home Telerehabilitation Program on Self-Care in Patients with Long COVID: a Randomized Clinical Trial
Brief Title: Effectiveness of a Personalized In-home Telerehabilitation Program on Self-Care in Patients with Long COVID
Acronym: RESPICARE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CEU San Pablo University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEU-028
Record Dates: First submitted 2025-02-11; First posted 2025-02-12 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Long COVID Syndrome
Keywords: post-acute COVID-19 syndrome; self-management; COVID-19; Rehabilitation; Exercise
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Motor Activity | interventions — Educational Status; Self-Management

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telerehabilitation program (Experimental): The interventions include:
  * Education for self-management
  * Personalised exercise program
  Interventions: Other: Education for self-management; Other: Personalised exercise program
- Control (Active Comparator): Usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Education for self-management — Education program performed online including information, recommendations and guidance for promoting self-management
  Arms: Telerehabilitation program
Other: Personalised exercise program — Individualized exercise that includes progressive load adapted to each patient. It includes making flexible adjustments to their exercise (up or down as needed) to help them gradually improve their physical abilities while staying within their energy limits
  Arms: Telerehabilitation program
Other: Usual Care — Usual care these patients may receive out from the clinical trial.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to evaluate whether a 12-week tele-rehabilitation programme with monitoring via a mobile app produces medium-term improvements in self-management, fatigue and quality of life in patients affected by persistent COVID.

The main questions it aims to answer are:

* Will a multimodal program (exercise with education) improve the self-management ability of patients with post-exertional malaise?
* Does fatigue and quality of life will be improved in these patients?

Researchers will compare an experimental breath program to a control standard care group to see if multimodal program works to treat post-exertion malaise.

Participants will:

* Follow-up 12 weeks online sessions:

  1 weekly synchronous online session + 1 scheduled asynchronous session + educational resources
* Daily use of the app: daily log, education and questions

ELIGIBILITY:
Inclusion Criteria:

* Post COVID-19 condition: individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis. Common symptoms include fatigue, shortness of breath, cognitive dysfunction
* Between 18 and 75 years of age
* Possibility of access and use of smartphone.
* Ability to attend the clinic in person for an initial session.

Exclusion Criteria:

* Patients with a history of respiratory or cardiovascular diseases prior to COVID-19, other acute or chronic diseases that may interfere with the study
* Pregnancy/breastfeeding
* Those with contraindications to respiratory muscle training.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Patient activation measure 13 | From enrollment to end of treatment and 3 months follow-up
  Individual's knowledge, skills and confidence to managing one's own health. is a non-disease-specific tool and can be used across different patient populations. The PAM-13 consists of 13 items on a 4-point Likert scale (1 = strongly disagree, 2 = disagree, 3 = agree, 4 = strongly agree). Item scores are summed up to a raw sum score resulting in theoretical values between 13 and 52, which are then transformed to a standardized metric ranging from 0 to 100. Higher scores indicate a greater patient activation. PAM-13 scores can then be categorized into four stages of activation, corresponding to the difficulty of the PAM-13 items: level 1 (patients believe active role is important; items 1-2), level 2 (patients have confidence and knowledge to take action; items 3-8), level 3 (taking action; items 9-11) and level 4 (staying on course under stress; items 12-13).
self-care self-efficacy scale | From enrollment to end of treatment and 3 months follow-up
  Measure for self-care self-efficacy for chronic illness. This 10-item instrument measures self-efficacy related to self-care maintenance, monitoring, and management in patients with chronic illness. Each item is rated on a '1-5' rating scale, with a higher score representing a higher level of self-efficacy. Scale scores are standardized mathematically to range from 0-100.

SECONDARY OUTCOMES:
Health-related quality of life EuroQol-5D | From enrollment to end of treatment and 3 months follow-up
  Quality of life related to dimensions of mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  Each dimension is described by three possible levels of problems (no, mild to moderate and severe). Hence, this descriptive system contains three or 243 combinations, or health states. For each of these combinations, one can assign healthstate utility indices (or ''preference weights'') which are based on different value sets.
Fatigue Severity Scale (FSS) | From enrollment to end of treatment and 3 months follow-up
  Severity of fatigue and its effect on a person's activities and lifestyle. The FSS questionnaire contains nine statements that rate the severity of your fatigue symptoms. Read each statement and circle a number from 1 to 7, based on how accurately it reflects your condition during the past week and the extent to which you agree or disagree that the statement applies to you. A low value (e.g., 1) indicates strong disagreement with the statement, whereas a high value (e.g., 7) indicates strong agreement. The minimum score=9 and maximum score possible=63. Higher the score=greater fatigue severity.
DePaul Symptom Questionnaire-Short Form (DSQ-SF) | From enrollment to end of treatment and 3 months follow-up
  The DSQ-SF allows investigators to use a small number of items (n = 14) to determine whether patients meet ME/CFS case definitions. Similar to the DSQ, the DSQ-SF uses the mean of the frequency and severity scores for each symptom rated over the past 6 months and linearly transforming it into a 100-point scale

CONTACTS AND LOCATIONS:
Locations (1):
- CEU San Pablo University, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No